CLINICAL TRIAL: NCT04416178
Title: Sickle Cell Disease and the Genomic and Gene Therapy Needs of Stakeholders
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: SCDGEN; 5U01HL133996 (NIH)
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Sickle Cell Anemia; Hemoglobin SC Disease; Hemoglobin SS Disease; Hemoglobin S beta zero thalassemia; Adolescent; Parent
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survey and Interview Group (Group1): Parent of child with HbSS, HbS/ β0thalassemia, β+ thalassemia or HbSC aged 12 months to 18 years at study initiation, irrespective of clinical severity or patient aged 13-18 with aforementioned SCD genotype.
- Usability and Pilot Testing (Group 2): Parent of child with HbSS, HbS/ β0thalassemia, β+ thalassemia or HbSC aged 12 months to 18 years at study initiation, irrespective of clinical severity or patient aged 13 and up with aforementioned SCD genotype.

SUMMARY:
The primary objectives of this prospective mixed-method interview study are to use semi-structured interviews in parents of sickle cell disease (SCD) patients to describe parental attitudes of research involving genomic sequencing, including concerns about participation and expectations from researchers and second, to use surveys to quantitatively measure genetic/genomic knowledge, trust in health care provider, and literacy/numeracy ability in parents of children with SCD and adolescents with SCD. Secondary objectives are development of a web-based tool about treatment options for SCD that fosters patient-clinician communication and promotes shared decision-making. The web-based tool will undergo usability and pilot testing to ensure it is accessible to families and provide data about strategies for integrating into clinical conversations about treatment options.

Investigators will use the data generated to reduce the risk of misunderstanding about DNA and genetic research and build strong relationships between SCD families and researchers in the future. The project will design educational information and study materials to help parents of children with SCD understand important details about genomic medicine in SCD care.

DETAILED DESCRIPTION:
There is a critical gap in knowledge regarding the attitudes, beliefs, and expectations of parents around clinical research trials involving genomic sequencing of children with sickle cell disease (SCD). SCD primarily affects children of African American (Black) race; institutionally we have found differences in enrollment on genomic sequencing trials (G4K (NCT02530658), PG4KDS) with patients identifying as black more likely to decline enrollment. Enrollment on SCCRIP (NCT02098863), a biobank study for children with SCD is high (92.3%), indicating that potential genomic research does not appear to concern many families with SCD. Given the rising prevalence of clinical research involving genomic sequencing in pediatric SCD, coupled with the increasing likelihood that sequencing will be required for enrollment on therapeutic drug or gene therapy trials, there is a clear need for research to better understand stakeholder concerns and expectations around genomic sequencing in this population.

Parents of children with SCD and adolescent patients will be approached to complete a short survey during a routine clinic visit, in the medicine room or in-patient. Survey questions will be administered at the time of the informed consent conversation. Those who agree will be given a paper survey or an ipad to complete survey items which focus on genetic/genomic knowledge, trust in health care provider, and literacy/numeracy ability in parents of children with SCD and adolescents with SCD. Participants also have the option to have questions read to them or they can take the survey on paper. Completion of the survey is expected to take < 30 minutes. Patient and parent can complete surveys simultaneously.

Of parents completing surveys, a subset will be approached for a private (in person or virtual) semi-structured interview. Participants willing to be interviewed will be interviewed at either the same study visit or at a future visit if this is more convenient for the participant. The interview guide (member of the study team) will ask questions designed to first assess parental perceptions about clinical research then begin to focus on parental attitudes, beliefs, and expectations around research involving clinical genomics. Interviews will be conducted on-site at St. Jude Children's Research Hospital in a private, quiet area. The interview should last 30-60 minutes and will be audio recorded. Some survey or interview study visits may occur remotely.

Investigators will re-approach 5-15 parents and 5-15 patients (both adolescent and young adult) to review educational materials developed about sickle cell disease treatment options. Additionally, investigators will approach parents of children with SCD as well as young adult patients for pilot testing of the web-based educational tool.

ELIGIBILITY:
Inclusion Criteria

Group 1 (Survey and Interview) Participants only:

* Parent of child with HbSS, HbS/ β0thalassemia, or HbSC aged 12 months to 18 years at study initiation, irrespective of clinical severity or patient aged 13-18 with aforementioned SCD genotype.
* Informed consent from parent or legal guardian and assent of adolescent participant.
* Has been previously approached for SCRIPP.

Group 2 (Usability and Pilot Testing) Participants only:

* Parent of child with HbSS, HbS/ β0thalassemia, β+ thalassemia or HbSC aged 12 months to 18 years at study initiation, irrespective of clinical severity or patient aged 13 and up with aforementioned SCD genotype.
* Informed consent from parent or legal guardian and assent of adolescent participant.

Exclusion Criteria (All groups):

* Participants who are unable to converse fluently in English will be excluded. (Permanent)
* Condition or chronic illness, which in the opinion of the PI/Co-I, makes participation unsafe or untenable (i.e. cognitive impairment, concurrent acute morbidity). Participant may be re-evaluated.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Those who meet the Eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Use of semi-structured interviews in parents of SCD patients to qualitatively describe parental attitudes of research involving genomic sequencing, including concerns about participation and expectations from researchers | Day 1, or at a future visit (up to approximately 1 year)
  Interviews will be audio recorded, transcribed verbatim and analyzed using semantic content analysis to identify common themes
Use of surveys to quantitatively measure genetic/genomic knowledge, trust in health care provider/researchers, and literacy/numeracy ability in parents of children with SCD and adolescents with SCD. | Day 1
  Patients and parents' demographic characteristics will be collected from the electronic medical record (EMR). Participants will complete various survey instruments designed to measure knowledge and attitudes around genetic testing and biobanks, self-reported literacy and numeracy, and trust in providers. Data will be analyzed quantitatively using descriptive statistics, generalized linear regression models and generalized estimation equations.

CONTACTS AND LOCATIONS:
Overall Officials: Liza M. Johnson, MD, MPH, MSB, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols